CLINICAL TRIAL: NCT00890877
Title: Dose Finding Study in Patients With Mild to Moderate Persistent Asthma: A Parallel Group, Randomised, Placebo Controlled, Double Blind Assessment of Oral Oc000459 Dosed At Three Dose Schedules for Twelve Weeks Finding Study In Patients With Mild To Moderate Persistent Asthma
Brief Title: OC000459 Dose Finding Study in Patients With Mild to Moderate Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxagen Ltd (Industry)
Responsible Party: Dr C Mike Perkins, Oxagen Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OC000459/012/08
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Mild to Moderate Persistent Asthma
Keywords: asthma; treatment; placebo; efficacy; safety
MeSH Terms: conditions — Asthma | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: OC000459 or placebo
- 2 (Experimental)
  Interventions: Drug: OC000459 or placebo
- 3 (Experimental)
  Interventions: Drug: OC000459 or placebo
- 4 (Experimental)
  Interventions: Drug: OC000459 or placebo

INTERVENTIONS:
Drug: OC000459 or placebo — Pills, active and/or placebo given twice daily for 17 weeks

SUMMARY:
This will be a double blind, randomised, 4 arm, parallel group, placebo controlled study of three dose levels of OC000459 tablets in patients with asthma controlled by beta agonist drugs alone. This study will compare the patients on OC000459 at three different dose levels (25mg once daily, 100mg twice daily and 200mg once daily) with patients on placebo after dosing for 17 weeks. The trial will be undertaken in an outpatient population. Each treatment arm will consist of at least 110 subjects. The objective is to assess the efficacy of these dose levels on the patients asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female asthmatics, any racial group. Females of childbearing potential must practise two forms of contraception
* Aged 18 to 55 years inclusive.
* Non smokers for at least the past 12 months with a pack history of less than 10 pack years.
* Mild to moderate persistent asthma according to GINA4 guidelines for at least 12 months

Exclusion criteria:

* Receipt of prescribed or over the counter medication within 14 days prior to the first study day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 17 weeks

SECONDARY OUTCOMES:
Asthma quality of life questionnaire (AQLQ) | 17 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Research site, Sofia, Bulgaria
- Research site, Győr, Hungary
- Research site, Warsaw, Poland
- Research site, Bucharest, Romania
- Research site, Moscow, Russia
- Research site, Kiev, Ukraine